CLINICAL TRIAL: NCT06820658
Title: A Comparison of Neuromuscular Recruitment in Trained and Untrained Adults
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, K. Sreekumaran Nair, Principal Investigator, Mayo Clinic
Other Study IDs: 21-000002; 1R01AG062859 (NIH)
Record Dates: First submitted 2025-01-21; First posted 2025-02-11 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Healthy; Insulin Resistance
Keywords: neuromuscular; transcranial magnetic stimulation
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Highly resistance-trained
  Interventions: Diagnostic Test: Neuromuscular Test; Diagnostic Test: DEXA; Diagnostic Test: Mixed Meal Tolerance Test; Diagnostic Test: Strength Test
- Untrained
  Interventions: Diagnostic Test: Neuromuscular Test; Diagnostic Test: DEXA; Diagnostic Test: Mixed Meal Tolerance Test; Diagnostic Test: Strength Test

INTERVENTIONS:
Diagnostic Test: Neuromuscular Test — To measure neuromuscular connectivity, Transcranial Magnetic Stimulation (TMS) will be used to stimulate regions of the cerebral cortex known to control specific muscles.
  Electromyography (EMG) activity will then be measured from the following muscle groups: deltoid, biceps, extensor digitorum communis, abductor pollicis brevis, abductor digiti minimi, and first dorsal interosseous muscle.
Diagnostic Test: DEXA — The DEXA test uses X-rays to measure how many grams of calcium and other bone minerals are packed into a segment of bone. The test also measures the amount of fat-free mass, and fat mass.
Diagnostic Test: Mixed Meal Tolerance Test — Fasting blood will be collected for glucose, insulin, and c-peptide. Participants will be provided with a milkshake with a fixed amount of protein, carbohydrates, and fat. Glucose, insulin, and c-peptide will be measured at multiple time points (every 10 minutes) until four hours after consumption (50% Fat, 30% Carbohydrate HO, 20% Protein). Approximately 70mls of blood will be drawn during this time
Diagnostic Test: Strength Test — Knee extensor strength will be tested by gradually increasing the workload on a pneumatic Keiser knee extension machine. The test will begin with a warm-up of 4-5 reps with one leg at 30-50 psi. Then the participant will increase the workload at self-selected intervals ranging from 5-20psi until a maximum effort is achieved. If a rep is failed, then the workload will be reduced by 5psi until a successful rep is performed or a workload is reached in which a successful rep had been previously achieved. Handgrip strength will be tested using a handheld dynamometer (Baseline® standard hydraulic hand dynamometer). The test is performed with the participant seated with the elbow unsupported and flexed at 90 degrees, forearm neutral, wrist held between 0-15 degrees of ulnar deviation (Horowitz, 1997). Maximum grip is the average of three 3-5 second trials.

SUMMARY:
The objective of the study is to use neurological techniques to obtain quantitative measurements of nervous system control of skeletal muscle activity in adults aged 60-85 who are either long-term resistance exercisers or who are untrained.

DETAILED DESCRIPTION:
We propose to perform a cross-sectional study in 20-40 highly resistance-trained people and compare with 20-40 untrained people matched for age, sex, and BMI. in adults.

Participant will complete 5 study visits. In the first visit, participants will complete a screening visit in which blood will be taken to rule out inclusion and exclusion criteria. Participants will also have their body composition measured by DEXA, Meal tolerance testing, a VO2max test on a cycle ergometer, and a muscle strength test using a knee extension machine, handgrip dynamometer and muscle motion testing.

A second and third visit will be needed for meal tolerance testing will be completed and MRI of the brain.

In the fourth and fifth visits, we will use transcranial magnetic stimulation (TMS) with electromyography (EMG) to track changes in in skeletal muscle excitability following cortical stimulation.

In the third visit, TMS-EMG measurements will be repeated to access measurement reproducibility.

ELIGIBILITY:
Inclusion Criteria

* Participant must have a BMI between 18.5 and 38
* Participant be aged between 60 and 85
* Regularly exercises at least 5 days a week a minimum of 30 minutes per day.
* Engages in less than 2 days of exercise less than 30 minutes each day.
* Participant must use the Mayo Clinic patient online portal.
* Participant must be able to understand English without the need of an interpreter.
* Must be willing to be contacted for research
* Participant must be willing and capable to provide consent.
* Participants shall be generally healthy as deemed acceptable by the principal investigator
* Men and women will be participant in this study. Women cannot be pregnant during this study.

Exclusion Criteria:

* Surgical History - Gastric surgery, pacemaker placement, weight loss surgery, metabolic and obstetric surgery.
* Smokers will be excluded from the study.
* Medications: Insulins, common diabetic drugs, anti-hyperglycemic drugs, beta blockers cardiac selective, beta-blockers noncardiac selective, oral steroids, opioids anti-depressants, and hormones
* Conidiations and Diagnosis: Disorder of coronary artery, hepatic failure, gastroparesis, disorder of the adrenal gland, drug related disorders, substance abuse, malignant neoplastic disease, psychotic disorders, disorder of skeletal muscle, finding of brain, chronic kidney disease, renal failure syndrome, disorder of pulmonary circulation, cerebrovascular disease, neuro developmental disorder, disorder of immune function, disorder of central nervous system.
* Participants are not to have an abnormal value as part of a lipid panel within the past 6 months.
* Participant will be excluded if they have recreational drug use or a history of alcohol abuse
* Inability or unwillingness of individual or legal guardian/representative to give written informed consent.
* Current or past participation within a specified timeframe in another clinical trial, as warranted by the administration of this intervention.
* Participant will be excluded if they have epilepsy.
* Participant will be excluded if they have cranial metal/device implants
* Participant will be excluded if they are pregnant

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 80 participants will be equally divided into resistance-trained and untrained groups. Participants will be matched for age, sex, and BMI. Participants are to have a fasting blood sugar under 140 mg/dL. Untrained men and women will have a hip to waist ratio of >0.85 in women or >80cm and >0.90 in men or >94cm. Participants will be from the Rochester Minnesota area aged 60-85 with a BMI 30-38.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Electromyography (EMG) response following Transcranial Magnetic Stimulation (TMS) | 21 days
  To assess connectivity between the nervous system and skeletal muscle, we will use transcranial magnetic stimulation (TMS) coupled with electromyography (EMG). TMS uses a magnetic field to carry a short-lasting electrical current pulse into the brain where it stimulates neurons, particularly in superficial regions of cerebral cortex, and neural activities can be measured at different levels along the motor pathways (predominantly the CST). When combined with EMG, this approach will allow us to quantify changes in muscular activity after stimulating the CST and other descending tracts and to assess the neuromuscular connectivity. EMG assess the health of muscles and the nerve cells that control them (motor neurons). EMG results can reveal nerve dysfunction, muscle dysfunction or problems with nerve-to-muscle signal transmission. Motor neurons transmit electrical signals that cause muscles to contract. Electrodes will then translate signals into graphs, sounds or numerical values.

CONTACTS AND LOCATIONS:
Overall Officials: K. S. Nair, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States